CLINICAL TRIAL: NCT00364325
Title: Acute Decompensate Heart Failure National Registry ( ADHERE) Emergency Module (EM)
Brief Title: Registry for Acute Decompensated Heart Failure Patients Admitted to the ER
Status: Completed | Type: Observational
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sr. Director, Clinical Team Leader, Scios
Other Study IDs: CR005215
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Heart Failure, Congestive; Heart Decompensation
Keywords: Heart failure, congestive; Heart decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Acute Decompensated Heart Failure

INTERVENTIONS:
Other: Acute Decompensated Heart Failure — Standard of Care

SUMMARY:
The purpose of this study is to collect data on the medical management of patients presenting to the Emergency Department who are treated for Acute Decompensated Heart Failure (ADHF) in a hospital setting that has incorporated a disease management program for heart failure.

DETAILED DESCRIPTION:
This is an Observational (individuals are observed or certain outcomes are measured. no attempt is made to affect the outcome), multi-center registry study of patients presenting to the Emergency Department (ED) for treatment of known or suspected Acute Decompensated Heart Failure (ADHF). Data will be collected on the medical management of patients presenting to the ED who are treated for ADHF in a hospital setting incorporating a disease management program for heart failure. The study will evaluate change in clinical management and outcomes of ADHF patients treated in the ED after ED implementation of three or more components of a disease management program for heart failure. The results are intended to assist hospitals in evaluating and improving quality of care for patients with ADHF by tracking quality indicators and providing site-specific benchmark reports and national benchmark reports. This registry considers patients treated with any therapy for ADHF

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of ED treatment
* Received or is eligible to receive a principal ED and/or hospital discharge diagnosis of ADHF
* ADHF is present as determined clinically by the patient care team and as documented in the DRG (Diagnosis-related Group) or APC (Ambulatory Payment Classifications) codes, and ADHF is the focus of treatment
* If required by site IRB/IEC patient (or legally acceptable representative) must be able to give informed consent for participation

Exclusion Criteria:

* ADHF is present as a co-morbid condition, but is not a principal focus of diagnosis or treatment during this ED or hospital episode
* Patient was not treated in ED during this episode of care
* Participation in any clinical trial that precludes use of a Disease Management Program (specific component of the disease are managed in an integrated manner by a team of physicians, pharmacists, nurses and communication experts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all consecutive adults patients seen in the Emergency department of an acute care hospital and treated actively for Acute Decompensated Heart Failure (ADHF) where the condition is defined clinically as new onset of Heart Failure with decompensation or chronic heart failure with decompensation. Patient eligibility is based upon the presence of a hospital discharge and/or Emergency department diagnosis of ADHF and is not tied to the use of any specific therapeutic agent or regimen.
Sampling Method: Non-Probability Sample
Enrollment: 18920 (Actual)
Dates: Start 2004-07; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The registry will capture information about the medical care that the patient has received including hospital/ emergency department course, major procedures, medication received, emergency room disposition and in hospital death | Data will be collected, beginning with care in the Emergency Department and ending with the patient's Discharge from the Emergency Department or hospital discharge, transfer to another hospital, or in-hospital death.

SECONDARY OUTCOMES:
Baseline demographic information (age,sex, gender,race), initial evaluation, laboratory results and medical history. | From admission to the emergency depatment until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.